CLINICAL TRIAL: NCT01834196
Title: Swept-Source Optical Coherence Tomography for Noninvasive Retinal Vascular Imaging
Acronym: SWEPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No active study enrollment for a 2 years.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00038240
Record Dates: First submitted 2013-04-15; First posted 2013-04-17 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2015-02

CONDITIONS: Retinal Vascular Disease
Keywords: retinal vascular disease; Swept-Source Ocular Coherence Tomography; SSOCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- retinal vascular occlusion arm (Other): Patients with existing retinal microvascular disease will undergo imaging.
  Interventions: Device: Swept-Source Optical Coherence Tomography

INTERVENTIONS:
Device: Swept-Source Optical Coherence Tomography — Noninvasive imaging of the retinal vasculature in patient with existing microvascular disease.

SUMMARY:
This is a clinical pilot study to assess the feasibility of using a swept-source optical coherence tomography (SSOCT) system to perform noninvasive imaging of the retinal vasculature in patients with existing microvascular disease.

DETAILED DESCRIPTION:
This project is being conducted under an abbreviated IDE. Subjects with existing retinal microvascular disease will be recruited from among the patients of the Duke Eye Center and/or its associated satellite clinics. Following informed consent, subjects undergo imaging, per established standard operating procedure, at the Duke University Medical Center/Duke Center or at one of the Duke Eye Center satellite clinics. Pharmacologic dilation of eyes will not be necessary for completion of imaging and will not be used for the purposes of this study. The resulting images will not be used in the clinical care of any of the subjects recruited for this project.

Subjects will be identified from patients presenting for ophthalmologic consultation at the Duke Eye Center and/or its satellite clinic locations.

ELIGIBILITY:
Inclusion Criteria:

1. Capable and willing to provide consent
2. history of clinically-diagnosed retinal microvascular diseases, including but not limited to diabetic retinopathy, retinal vein occlusion, idiopathic macular telangiectasias, hypertensive retinopathy, and age-related macular degeneration
3. At least 18 years of age

Exclusion Criteria:

1. Unable or unwilling to give consent
2. Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
OCT images and metrics derived from the OCT images | Day of imaging, approximately 1 hour
  Distributions, means, and standard deviations will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Prithu Mettu, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States